CLINICAL TRIAL: NCT05605028
Title: PowerObesity: Community Lifestyle Interventions to Prevent and Improve Mental Health of Minorities
Brief Title: A Mental Health Intervention for a Community Program Called the PowerObesity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: I needed it to have the position of professor at the university and by the time the professorship was given it was too late for the grant therefore there is no funding and the study was never started.
Sponsor: Charles Drew University of Medicine and Science (Other)
Responsible Party: Principal Investigator, Eddie Ramirez, Research Assistant Professor, Charles Drew University of Medicine and Science
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Mental Health for PowerObesity
Record Dates: First submitted 2022-10-18; First posted 2022-11-03 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Mental Health Wellness 1; Depression; Anxiety; Sedentary Behavior; Obesity; Poor Nutrition
MeSH Terms: conditions — Depression; Anxiety Disorders; Sedentary Behavior; Obesity; Malnutrition

STUDY DESIGN:
Intervention Model Description: The intervention will take 1 year to recruit all the patients. The investigators expect to have the 75 patients in the group intervention and 25 patients in the dietitian-led group. With these numbers, our preliminary power analysis suggests there will be a difference in the two groups with an alpha of .05 and 80% power. The investigators will add 3 tests to both arms of the study, 9-question Patient Health Questionnaire (PQ-9), Generalized Anxiety Disorder (GAD), and the Depression and Anxiety Assessment Test, in the POWER Obesity group at 0, 3, 6 months and 12 months of intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Health lifestyle intervention (Experimental): The intervention will focus on identifying risk factors for depression and anxiety and will quantitate the educational component of the POWER Obesity group intervention delivered by mental health professionals that are currently presenting for 30 min during the Monday session to address the root causes of obesity as well as to encourage positive lifestyle changes (e.g. sleep, diet, sun exposure, circadian rhythms, and addictions). The previously published hypothesis identifies triggers, that combined, could cause mental health problems. The 10 groups of triggers are: (1) Genetic, (2) Developmental, (3) Lifestyle, (4) Circadian Rhythm, (5) Addiction, (6) Nutrition, (7) Toxic, (8) Social/Complicated Grief, (9) Medical Condition, and (10) Frontal Lobe. Each of these factors will be dealt with in the lifestyle intervention.
  Interventions: Behavioral: Mental Health lifestyle intervention
- Dietitian-led (Active Comparator): A group of participants that visit a dietitian will be the control.
  Interventions: Other: Dietitian-led

INTERVENTIONS:
Behavioral: Mental Health lifestyle intervention — The focus is to identify 10 potential groups of causes and working on reversing them. The 10 factors are: (1) Genetic, (2) Developmental, (3) Lifestyle, (4) Circadian Rhythm, (5) Addiction, (6) Nutrition, (7) Toxic, (8) Social/Complicated Grief, (9) Medical Condition, and (10) Frontal Lobe. Each of these factors will be dealt with in the lifestyle intervention.
  Other Names: 10 hit hypothesis intervention
  Arms: Mental Health lifestyle intervention
Other: Dietitian-led — A group of people that visit the dietitian will be used as comparison against the Mental Health lifestyle intervention
  Arms: Dietitian-led

SUMMARY:
The intervention will focus on identifying risk factors for depression and anxiety and will quantitate the educational component of the POWER Obesity group intervention delivered by mental health professionals that are currently presenting for 30 min during the Monday session to address the root causes of obesity as well as to encourage positive lifestyle changes (e.g. sleep, diet, sun exposure, circadian rhythms, and addictions). The previously published hypothesis identifies triggers, that combined, could cause mental health problems. The 10 groups of triggers are: (1) Genetic, (2) Developmental, (3) Lifestyle, (4) Circadian Rhythm, (5) Addiction, (6) Nutrition, (7) Toxic, (8) Social/Complicated Grief, (9) Medical Condition, and (10) Frontal Lobe. Each of these factors will be dealt with in the lifestyle intervention. The project will be led by the assistant professor (in process) Francisco E Ramirez, MD with his mentor Theodore Friedman, MD, PhD supervising the project.

Hypothesis:

The investigators hypothesize that composite POWER Obesity group will have greater improvement in mental health compared to the dietitian-led group.

Measuring outcomes:

The intervention will take 1 year to recruit all the patients the investigators expect to have the 75 patients in the group intervention and 25 patients in the dietitian-led group. With these numbers, our preliminary power analysis suggests there will be a difference in the two groups with an alpha of .05 and 80% power. The investigators will add 3 tests to both arms of the study, 9-question Patient Health Questionnaire (PQ-9), Generalized Anxiety Disorder (GAD), and the Depression and Anxiety Assessment Test, in the POWER Obesity group at 0, 3, 6 months and 12 months of intervention.

DETAILED DESCRIPTION:
Research plan A. Significance A.1 Rationale The obesity epidemic in the north American population is a growing concern amongst the scientific community. Diabetes and cardiovascular disease have been shown to be significantly influenced by obesity. The Centers for Disease Control and Prevention (CDC) defines obesity as having a body mass index (BMI) greater than or equal to 30 m/kg2, which is determined by a person's height and weight. A recently published systematic analysis of body mass index in 199 countries and territories showed a trending increase in the BMI of individuals in the United States alone from 1980 to 2008, ranking the highest in both male and female BMI ranges for high income countries . The United States also ranked the highest for obesity rates (23.9%) in a study analyzing possible correlations between obesity and active transportation in Europe, North America, and Australia . In addition, a study looking at the overall increasing trend of obesity in America estimated that with the current annual progression of obesity rates in America, that 86.3% of adults will be obese by 2030 . Women of non-Hispanic African descent are 56.7% obese, while Latinas are 44.4% obese . There is a need for affordable health programs that could available to the general population. Another program facing the community in the area of study is mental health problems. According to the World Health Organization, depression is "the leading cause of disability worldwide" and "a major contributor to the overall global burden of disease" . This accumulating problem leads many towards dysfunction, decreased efficiency, loss in quality health, increased addictive behaviors, and even suicide. Also, studies show that major depression and alcohol dependence were "associated with heavy cigarette use and poor smoking-treatment outcomes . In their study the investigators demonstrated that programs that improve overall health can also improve mental health , .

A facilitated lifestyle-based program like the Complete Health Improvement Program (CHIP) has been shown to help lose weight, lower their risks of heart disease and mental health . Through a balanced approach, program participants are instructed on how to make healthier food choices, incorporate regular physical activity into their daily lives, learn stress management techniques, and stop using tobacco (if applicable).

A.2 Can a lifestyle education program work for mental health and obesity? Community education programs that deal with the root causes of the problems are very effective in changing behavior and improving overall health . Some of the root issues with obesity and mental health. The program focuses on improving lifestyle of participants. These are some of the lifestyle interventions that will be used and their effectiveness.

Healthy diet Healthy lifestyles involve eating a balanced diet, maintaining a healthy weight, working out regularly, being low to moderately stressed, not smoking, and limiting alcohol consumption. A healthy diet has been proven to lower the risk of heart disease. The Mediterranean Diet, for instance, has been shown to lower heart disease risk by up to 70% compared to dieting alone . In addition, nearly half of the money Americans spend on food is spent at fast-food restaurants, which is double what was spent in 1955 . Fat, sugar, and salt are typically high in restaurant meals, which can contribute to heart disease. found that a healthy diet contains a balance of essential nutrients, calories, carbohydrates, fats, and protein, which reduces the risk of heart disease .

Reducing body weight An additional contributor to these diseases is obesity. The effects of obesity on cardiovascular disease and diabetes have been well documented. Obese individuals are at risk for a variety of health issues, including high cholesterol, diabetes, hypertension, heart disease, and stroke . Coronary heart disease, also known as coronary artery disease, is one of the deadliest health issues associated with obesity. The National Institutes of Health (NIH) reports that your arteries can become narrow as a result of fat, cholesterol, and calcium building up and forming plaque in your arteries . Angina, shortness of breath, and arrhythmia are some of the signs and symptoms of coronary heart disease.

* Exercise 150 minutes of moderate intensity physical activity per week can improve cholesterol levels . In the intervention the investigators are proposing, physical activity recommendations serve as guidelines improve overall health. Physical activity rates and obesity rates among Americans emphasize the importance of focusing on fitness and weight management. The American Heart Association reports that only 49.1% of American adults met the recommended physical activity standards . The Centers for Disease Control and Prevention (CDC) data show that 24.1% of American adults did not participate in leisure-time physical activity that same year. Compared to 1950, the number of sedentary occupations has increased by 83%, while the number of physically active jobs has decreased by 25% , .
* Control of stress Mental health, obesity and other problems are also associated with stress. A person's heart rate and blood pressure increase when they are faced with a stressful situation . There is also evidence that individuals suffering from anxiety, depression, and anger are more likely to develop heart disease . When examining current American lifestyles, which are characterized by chronic stress, this information can be cause for concern. Therefore, Americans may be at increased risk for multiple health problems. Furthermore, many Americans find it difficult to balance work, finances, family life, and time to practice healthy habits .

A.3 Nutrition therapy Dietitians (RDs) and nutritionists (RDNs) provide food and nutrition education as well as medical nutrition therapy . In both short- and long-term studies and in both group and individual settings, Micronutrient test (MNT) administered by a RD or RDN is associated with significant weight loss both statistically and clinically. Dietitian-led individualized visits provide a control for the study.

A.4 Medical Group visits The group visit is not the same as a class or group therapy session and clearly differs from other for-profit models which do not address health disparities directly or mitigate them. These models have been used to conduct group visit programs for a variety of medical conditions in multiple practice settings , . When compared with standard individual medical visits, medical group visits have been shown to be associated with clinically significant improvements in a variety of medical, psychological, and behavioral outcomes , , . Medical group and high-risk populations, such as elderly patients , medical group visits have proven to be highly effective methods for improving access to medical care and monitoring complex chronic diseases. The utilization of emergency departments and outpatient services is decreased in patients treated through medical group visits, their quality-of-life increases, and their satisfaction with their care is higher .

A.5 Gaps in evidence in treating depression Depression is usually treated in primary care settings using pharmacotherapy and psychotherapy as mainstays of treatment. Most patients with depression are treated by their primary care provider; approximately 5% to 10% of all patients at primary care clinics receive depression treatment . In almost 90% of cases, clinicians recommend antidepressant medications alone or in conjunction with psychotherapy to their patients who are diagnosed as suffering from depression . Antidepressants are currently the most prescribed class of medication in the U.S. , . Such medications as serotonin reuptake inhibitors, monoamine oxidase inhibitors, tricyclic antidepressants, and other atypical formulations target the dysregulation of neurotransmitters found in depression . Chronic illnesses, including depression, can be influenced by lifestyle and environmental factors, which are often overlooked. Researchers estimate that up to 80% of chronic diseases, such as heart disease, stroke, and diabetes, are caused by lifestyle choices and environmental factors , . A substantial portion of the variance in susceptibility to chronic diseases can be attributed to lifestyle factors and environmental factors , . Poor nutrition, physical inactivity, poor sleep hygiene, unmanaged stress, social isolation, and substance abuse are some examples , . Lifestyle medicine focuses on modifying these maladaptive lifestyle behaviors. The American College of Lifestyle Medicine defines lifestyle medicine as an evidence-based medical practice that promotes health and well-being through evidence-based therapeutic lifestyle modalities .

Positive lifestyle changes can reduce depression in several ways. The Mediterranean diet, which incorporates a higher intake of fruits and vegetables, has been associated with a decreased risk of depression . Studies have shown that moderate exercise of 20 minutes per day, 3 times per week can help reduce depression symptoms . Sleep hygiene interventions have been shown to reduce depression symptoms without pharmacological interventions . Active leisure can contribute to better mental health, especially for those who are unemployed, by increasing their perception of spending their time efficiently and effectively . Evidence-based training can help relieve mood disorders such as anxiety and depression , . Intimate and supportive relationships with family, friends, or significant others have been shown to be beneficial to mental health . Individuals who feel as though their lives have meaning tend to manifest fewer symptoms of depression .

A.6 10 hit hypothesis approach to mental health improvement The intervention will focus on identifying risk factors for depression and anxiety and will quantitate the educational component of the intervention delivered by mental health professionals that are currently presenting for 30 min during the Monday session to address the root causes as well as to encourage positive lifestyle changes (e.g. sleep, diet, sun exposure, circadian rhythms, and addictions). The previously published hypothesis . The hypothesis proposed by Nedley and Ramirez identifies triggers, that combined, could cause mental health problems. The 10 groups of triggers are: (1) Genetic, (2) Developmental, (3) Lifestyle, (4) Circadian Rhythm, (5) Addiction, (6) Nutrition, (7) Toxic, (8) Social/Complicated Grief, (9) Medical Condition, and (10) Frontal Lobe. Each of these factors will be dealt with in the lifestyle intervention.

B. Innovation The innovating proposal is to use medical group visit to encourage positive lifestyle changes that not only will have an impact on weight control but also on mental health in which the minorities around the institution will benefit. The control group will be a dietitian led program that provides obesity care for the inner-city population. The investigators will measure depression and anxiety as well as try to identify causes of depression and anxiety to encourage people to do the changes proposed. By the help of this Accelerating Excellence in Translational Science (AXIS) grant the investigators will be able to help the Los Angeles County (LAC)-Department of Health Services (DHS) population. This approach if successful could be replicated to improve obesity and mental health care in a sustainable way that could impact many people.

C. Approach C.1a Martin Luther King (MLK) POWER obesity group visit Endocrinologist Dr. Theodore Friedman (PI) and colleagues at the Martin Luther King Jr. Multi-Service Ambulatory Care Center (MLK MACC) [the name of the center changed to Martin Luther King Jr. Outpatient Center (MLK OC)] began providing obesity group visits in January 2013. The clinic, named POWER (Preventing Obesity With Eating Right), is open weekly on Monday afternoons for about 2 1/2 hours and patients can attend weekly or monthly. In 2014, the investigators changed the format to have English sessions on the 1st, 2nd and 5th Mondays and Spanish sessions on the 2nd and 4h Mondays. University of California, Los Angeles (UCLA) Clinical and Translational Research Institute (CTSI) provided funding to the Charles R. Drew University (CDU) through a research infrastructure grant, of which CDU is an equal partner. Using the preliminary funding, the investigators were able to obtain CDU Institutional Review Boards (IRB) approval, set up a database to track patients, hire a part-time coordinator, and increase the number of patients who attended clinics in person and via video conferencing. The investigators were able to set up an infrastructure for the proposed study through the pilot funding, allowing us to start recruiting patients for the pragmatic study immediately following funding. Power analysis can also be based on the data collected.

Our current POWER group visit at MLK begins with registration, vital signs, and 20 minutes of fitness. In this period, new subjects are informed they are part of an IRB-approved study that collects and anonymizes their data. Participants in the study are consented by the study coordinator (90% have consented). In a 30-minute overview, Dr. Friedman or another expert discusses the differences between diet and long-term lifestyle changes focusing on the complications of uncontrolled obesity and the benefits of weight loss, the importance of a plant-based diet, and physical activity. Each participant is then given a physical activity "prescription", both aerobic and strength training, on a prescription pad. Providers from orthopedics, mental health, and dentistry are frequent guest lecturers who discuss how obesity affects their fields. This visit concludes with a lecture by our dietitian using the curriculum. "Instant Recess" (which incorporates physical activity breaks into the daily routine to boost health and productivity) is discussed and our dietitian offers a lecture based on the curriculum. During the meeting, individuals are encouraged to ask lots of questions and to discuss their successes and barriers with the physician and with one another. The sessions last about 2 1/2 hours, and surveys indicate that participants are satisfied with the length and duration of the program. Each visit follows a standardized format. There are, however, updates to the slides and a variety of topics are discussed so that patients can get new information at subsequent appointments. On October 8, 2013, the Spanish language television station Univision profiled the obesity group visit program on its front page. The fitness was included in the visit in January 2011 and was highlighted on both the Channel ABC7 evening news and Univision evening news on August 10, 2015.

C.1b Pilot study The Power Clinic pilot IRB was approved in October 2013, 651 patients consented for that pilot program. Most of patients had diabetes or prediabetes. Regarding weight lost 30% of them lost at least 8 pounds. 12% lost at least 5% of their weight. Those who came more often showed better results. Most participants were satisfied with their experience and results. Input was taken from the patients, and they wanted the program to continue, the investigators also took many of their comments and improved the program overall.

As a result, our preliminary data indicates a solid infrastructure, recruitability, and success. Thus, the investigators are in a good position to implement the mental health proposal as soon as it is funded, the investigators only need a CDU IRB amendment for its approval.

C 1.c Mental health component. The mental health component to the intervention will be based on the 10 hit hypothesis. That approach has more than 80 presented abstract in various scientific meetings showing the effectiveness of applying lifestyle interventions , .

C.2 Study Design and approach. The investigators will do a randomization of the participants for the 18 months comparing those seeing a dietitian and those that will be learning about the 10-hit hypothesis. The study will randomize 75 participants with a 3:1 block ratio goal. By increasing the number of participants in the intervention group of the novel approach to mental health and to decrease the load of the dietitian led group. Participants can't choose which group to belong in order to improve the randomization of the trial. Patients cannot be in both arms of the study.

The recruitment method will be the same that was used to get the current Power Obesity group. The investigators will invite patients from obesity group to this sub study. Every patient that wants to participate of this mental health component need to consent. Both arms of the study are evidenced based the investigators will have minimum risk. If a participant does not want to consent, the investigators will provide them with a list of other options for them to benefit.

The group visits, 2 and a half days will be in Spanish and 2 and a half group will be in English. Each visit 2 ½ hours. For the dietician group of the study the intervention will be offered in English and Spanish. Participants can participate of the program if they want. The investigators will use 12 months of data for the study. Los Angeles county will benefit from both legs of the study of this cost-effective approach.

C.3.a Approach of both study arms.

The emphasis of the Power Obesity is to promote healthy behaviors: a) decrease refined foods. B) decreased consumption of simple refined carbohydrates c) decrease sugary beverages d) a goal of 150 min of aerobic exercise and 30 minutes of anaerobic exercise. Both groups will be assessed by the:

the International Physical Activity Questionnaire (IPAQ) which assessed the amount of exercise the participant does.

C 3.b Composite group visit. It will have all the element of the visit. 1) a lecture by an expert, 2) Guided exercise, 3) exercise prescription, delivery of the curriculum outlined by the National Diabetes Prevention Program. The visits will be documented in medical records in a system call ORCHID. The duration is going to be 2 ½ hours. The intervention will be offered in Spanish and English. In addition to the usual curriculum the mental health component. The mental health presentation will cover various areas from defining depression and anxiety, to what contributes to it, to who is at risk for these disorders and if recovery is possible. The investigators will have share for 20 minutes an evidenced based mental health component. Participants will be encouraged to adequately hydration, listen to more music therapy, begin or continue a good exercise program, and develop a more intentional way of thinking by listing things that they are grateful for. It will also deal with signs and symptoms of anxiety and various lifestyle therapies such as deep breathing, light therapy, exercise, and avoiding pessimistic thinking to combat depression and anxiety. Improving brain health through proper nutrition. A whole food, plant-based diet will be encouraged. Intake of omega-3 fatty acids will recommend as well as enough tryptophan and other vitamins and minerals from their foods. The person's thinking process on depression and anxiety. The benefits of cognitive behavioral therapy and correct thinking were presented along with various remedies for distorted thinking patterns. Addictions will be addressed in the program. Various addictions that can lead to depression or anxiety will be dealt with, two of them being alcohol and narcotics. Those with severe alcohol or benzodiazepine addictions will be encouraged to see a health professional. The common characteristics of addictions with the need to overcome addictions. The investigators will also deal with principles of cognitive behavioral therapy strategies, dealing with loneliness and grief, overcoming loss, and enhancing the frontal lobe function.

An accountability checklist will be used with each participant to complete daily. The checklist include accounting for water intake, omega-3 fatty acid intake, and proper amount of exercise, etc. The participants bring the checklist to every session to show that the tasks in each category were accomplished. The checklist will be utilized to encourage compliance with the things that were taught .

C 3.c Dietitian led visit This will follow the Academy of Nutrition and Dietetics guidelines . An individualized plan will be presented to each of the participants. It will last 1 hour each appointment will follow up appointment of 30 minutes. The focus will be in evaluating caloric intake, increase physical activity and other behavior changes with the goal of achieving a 10% weight loss from baseline.

C 3.d Inclusion criteria Age 18+, BMI more than 30 kg/m2, that want to lose weight. Currently eligible or currently able to receive care at the LAC-DHS a physician willing to adjust their medications. If patients are taking weight loss medication like orlistat, lorcaserin, and phentermine/topiramate-ER, phenetermine, diethylpropion, phendimetrazine and benzphetamine they could enroll if they stop the medication 2 months or more before joining. If they take a weight loss supplement, they need to stop it 3 months before participating. The investigators exclude pregnant participants due to the difficulty of tracking their weight. Those with bariatric surgery will be able to enroll if the surgery was 1 year before joining.

C 3e Recruitment strategy LAC-DHS and its community partners will recruit patients primarily. There are four medical centers and 19 clinics in LAC-DHS, and many of them have patient-centered medical homes (PCMH) and other primary care clinics. Among the community partners is the Southside Coalition of Community Health Centers, which consists of 8 clinics that can refer patients to LAC-DHS for specialty care, including obesity care. In their 15-20-minute visits, primary care providers in LAC-DHS usually do not have time to address lifestyle changes for obese patients and may refer them to a dietitian or obesity program (such as the POWER obesity clinic at MLK OC). With the introduction of eConsults (a DHS-wide platform that allows PCPs to refer patients to specialists for specialized care, including obesity treatment), LAC-DHS has improved communication among providers. Within LAC-DHS, there are about 200,000 obese patients. All primary providers can arrange a remote consultation with specialists through the eConsult portal, where the obesity clinic and study information can be found. The DHS Endocrinology Work Group, in which endocrinologists from all the medical centers meet biweekly to discuss endocrinology issues, is chaired by Dr. Friedman. An excellent way to disseminate information about the obesity group clinics and the study. Moreover, word-of-mouth referrals and advocacy from our patients in the obesity program will also increase. Los Angeles County Department of Health Services provides care to low-income Medicare beneficiaries (Covered CA) as well as patients without insurance. In ORCHID, visits are tracked by a "visit charge" that is not charged to patients.

A high percentage of Hispanics and African Americans is expected to participate. Native Americans, Pacific Islanders, those with substance abuse histories, as well as individuals with mental illnesses and disabilities may be recruited. Despite their low representation in the general population, the investigators expect to recruit Caucasians. Covariant analyses will be conducted on the major ethnic/racial groups.

C.3 Specific Aim 2 study design and approach. The intervention will aim to recruit the 75 participants for the group intervention and 25 participants for the dietitian-led group. With these numbers, our preliminary power analysis suggests there will be a difference in the two groups with an alpha of .05 and 80% power.

C 3.a Measures For this intervention. The investigators will add 3 tests, in addition to those tests already given at Power Obesity, to both arms of the study, 9-question Patient Health Questionnaire (PQ-9), Generalized Anxiety Disorder scale (GAD), and the Depression and Anxiety Assessment Test, at 0, 3 months, 6 months and 12 months of intervention.

E. Expected outcomes Although it is difficult to predict weight loss, based on our experience so far, the investigators expect approximately 5% of patients to lose over 10 pounds and another 10% to lose over 5 pounds during the course of the program. Another 35% should lose between 2-5% of their weight and the remaining 50% should not lose any weight (although their education and lifestyle will likely improve). Improved mental health markers are expected, as well as better International Physical Activity Questionnaire (IPAQ) scores and the healthy eating index.

Recruiting/consenting goals are realistic. Since LAC-DHS will be recruiting from all parts of the region, the recruitment goals are quite attainable. With the assistance of two volunteer students, the investigators recruited 434 patients in 34 months in the past, with Ms. Duran as the study coordinator dedicating 25% of her time to the project. As a study coordinator, she will recruit student interns. In terms of recruiting participants and completing the study, the investigators do not expect to have any difficulties. One of the strengths of our proposal is the diversity of the participants, but one of its limitations may be the lack of Caucasians and middle and upper class participants. In our view, this is only a minor limitation, as most studies under-represent minorities and treatment programs for safety net clinics must be cost-effective and pragmatic.

F. Sustainability:

Since the resources of LAC-DHS are being used the investigators expect the program to continue improving and even expand once the program finishes.

One of our main goals is to published multiple studies in order to inspire others to replicate the model and help many. The investigators plan to do this regardless of the outcomes.

G. Future direction Our study will end up answering many of our baseline questions and at the same time it will be creating new questions to be answered in the future. The study has a potential to be expended with bigger samples and other sites. The results of the study will determine which direction the study will go.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 or older,
* BMI > 30 kg/m2
* Open to either being part of a group visit or being coached by a dietitian.
* Must be currently receiving care at LAC-DHS or be eligible for this care and be enrolled in a primary care provider (PCP) capable of adjusting their medicines, including anti-hypertensive and diabetic medications,
* It is not necessary to have diabetes or hypertension in addition to obesity to enroll.

Exclusion Criteria:

* Currently participating of an obesity treatment program
* Currently taking weight loss medications such as orlistat, lorcaserin, phentermine/topiramate-ER, phenetermine, diethylpropion, phendimetrazine, and benzphetamine They can enroll if they have stopped taking weight loss medicine for at least two months.
* Those actively suicidal.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-02 (Estimated); Primary Completion 2025-12-02 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PQ-9) Test | Taken at baseline.
  Measures depression using Patient Health Questionnaire (PQ-9). Total score ranges from 0 to 27. The higher the score means a worse outcome.
Patient Health Questionnaire (PQ-9) Test | Taken at 3 months of intervention
  Measures depression using Patient Health Questionnaire (PQ-9). Total score ranges from 0 to 27. The higher the score means a worse outcome.
Patient Health Questionnaire (PQ-9) Test | Taken at 6 months of intervention
  Measures depression using Patient Health Questionnaire (PQ-9). Total score ranges from 0 to 27. The higher the score means a worse outcome.
Patient Health Questionnaire (PQ-9) Test | Taken at 12 months of intervention
  Measures depression using Patient Health Questionnaire (PQ-9). Total score ranges from 0 to 27. The higher the score means a worse outcome.
Generalized Anxiety Disorder (GAD-7) Test | Taken at baseline
  Measures depression using the Generalized Anxiety Disorder (GAD-7). Total score ranges from 0 to 21. The higher the score means a worse outcome.
Generalized Anxiety Disorder (GAD-7) Test | Taken at 3 months of intervention
  Measures depression using the Generalized Anxiety Disorder (GAD-7). Total score ranges from 0 to 21. The higher the score means a worse outcome.
Generalized Anxiety Disorder (GAD-7) Test | Taken at 6 months of intervention
  Measures depression using the Generalized Anxiety Disorder (GAD-7). Total score ranges from 0 to 21. The higher the score means a worse outcome.
Generalized Anxiety Disorder (GAD-7) Test | Taken at 12 months of intervention
  Measures depression using the Generalized Anxiety Disorder (GAD-7). Total score ranges from 0 to 21. The higher the score means a worse outcome.
Depression and Anxiety Assessment Test | Taken at baseline
  Measures depression and causes of depression using the Depression and Anxiety . Assessment Test. It reports which of 10 possible triggers of depression the patient has at the moment the test was taken. The text triggers are: Genetic, Developmental, Lifestyle, Circadian Rhythm, Addiction, Nutrition, Toxic, Social/Complicated Grief, Medical Condition, and Frontal Lobe.
Depression and Anxiety Assessment Test | Taken at 3 months of intervention
  Measures depression and causes of depression using the Depression and Anxiety . Assessment Test. It reports which of 10 possible triggers of depression the patient has at the moment the test was taken. The text triggers are: Genetic, Developmental, Lifestyle, Circadian Rhythm, Addiction, Nutrition, Toxic, Social/Complicated Grief, Medical Condition, and Frontal Lobe.
Depression and Anxiety Assessment Test | Taken at 6 months of intervention
  Measures depression and causes of depression using the Depression and Anxiety . Assessment Test. It reports which of 10 possible triggers of depression the patient has at the moment the test was taken. The text triggers are: Genetic, Developmental, Lifestyle, Circadian Rhythm, Addiction, Nutrition, Toxic, Social/Complicated Grief, Medical Condition, and Frontal Lobe.
Depression and Anxiety Assessment Test | Taken at 12 months of intervention
  Measures depression and causes of depression using the Depression and Anxiety . Assessment Test. It reports which of 10 possible triggers of depression the patient has at the moment the test was taken. The text triggers are: Genetic, Developmental, Lifestyle, Circadian Rhythm, Addiction, Nutrition, Toxic, Social/Complicated Grief, Medical Condition, and Frontal Lobe.

IPD SHARING:
Plan to Share IPD: Undecided
By the end of the intervention the investigators will make the decision.

REFERENCES:
- [Background] Nedley N, Ramirez FE. Nedley Depression Hit Hypothesis: Identifying Depression and Its Causes. Am J Lifestyle Med. 2016 Nov;10(6):422-428. doi: 10.1177/1559827614550779. Epub 2014 Nov 10. PMID 27885322